CLINICAL TRIAL: NCT07203534
Title: The Effect of Virtual Reality Headsets on Pain and Anxiety in the Peri and Post Bone Marrow Biopsy Period
Brief Title: ONC-MM-2407: The Effect of Virtual Reality Headsets on Pain and Anxiety in the Peri and Post Bone Marrow Biopsy Period
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00136466; ONC-MM-2407 (Other: Atrium Health); P30CA012197 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancy
Keywords: Bone Marrow Biopsy; Virtual Reality Headset
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other)
  Interventions: Other: Standard of Care
- Virtual Reality intervention and Standard of Care (Other)
  Interventions: Other: Standard of Care; Other: Virtual Reality intervention

INTERVENTIONS:
Other: Standard of Care — Standard of care for a bone marrow biopsy/bone marrow aspiration includes routine site-specific lidocaine anesthetic.
Other: Virtual Reality intervention — Participants will wear the VR headset (Quest 3 by Meta) during your bone marrow procedure.
  Arms: Virtual Reality intervention and Standard of Care

SUMMARY:
The purpose of this research study is to see if a virtual reality (VR) headset is useful in reducing physical discomfort and anxiety experienced by patients who are scheduled to undergo a bone marrow biopsy (BMB) and/or bone marrow aspiration (BMA).

DETAILED DESCRIPTION:
This will be a randomized controlled trial comparing standard of care to standard of care + VR intervention for adult participants who have or are suspected of having a malignant hematologic disorder and are scheduled for an outpatient bone marrow biopsy (BMB) and/or bone marrow aspiration (BMA). Participants will be randomized 1:1. Participants will be risk stratified based on whether they are undergoing a biopsy for the first time or not.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an IRB-approved informed consent directly.
2. Must be 18 years or older at time of consent.
3. Scheduled for an outpatient bone marrow biopsy (BMB) and/or bone marrow aspiration (BMA). Note that this does not need to be the participant's first BMB/BMA.
4. Participant should be suspected of or being diagnosed with a malignant hematologic disease (i.e., Acute or chronic leukemia, lymphoma, clonal plasma cell disorder, etc.) per the investigator.
5. Ability to read and understand the English language.
6. As determined by the enrolling investigator, ability of the participant to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Participant is prescribed analgesics or anxiolytics for the purpose of reducing pain or anxiety prior to the procedure.
2. Participant with known intolerance to using virtual reality devices, significant motion sickness, history of seizures, history of vestibular disorders, or heart conditions (unstable angina, recent myocardial infarction within the last 3 months, decompensated heart failure, uncontrolled arrhythmias-ventricular tachycardia, a fibrillation with rapid ventricular rate), history of postural orthostatic tachycardia syndrome (POTS) per participant report.
3. Participants with pacemakers, defibrillators, hearing aid, or other implanted medical device. The Meta Quest device contains magnets and components that emit magnetic/electromagnetic fields which could affect the operation of nearby electronics and medical devices.
4. Planned to undergo the bone marrow biopsy/bone marrow aspiration via Interventional Radiology or as an inpatient admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale Pain Scores Immediately Post-biopsy | Single time point evaluation completed immediately following biopsy procedure
  For each participant, the Numeric Rating Scale (NRS) score immediately post-biopsy will be captured indicating the participants' severity of pain. The score for each participant will be categorized into 6 ordinal categories (0 No Pain, 1-2 Very Mild, 3-4 Mild, 5-6 Moderate, 7-8 Severe, 9-10 Unbearable) and used to assess if those using the Virtual Reality Headset during the procedure experienced less overall pain immediately following the bone marrow biopsy.

SECONDARY OUTCOMES:
Single time point evaluation completed immediately following biopsy procedure | Single time point evaluation completed 24 hours after biopsy procedure.
  For each participant, the Numeric Rating Scale (NRS) score 24 hrs (-6 hrs/+12 hrs) post-biopsy will be captured indicating the participants' severity of pain. The score for each participant will be categorized into 6 ordinal categories (0 No Pain, 1-2 Very Mild, 3-4 Mild, 5-6 Moderate, 7-8 Severe, 9-10 Unbearable) and used to assess if those using the Virtual Reality Headset during the procedure experienced less overall persisting pain.
State Trait Anxiety Inventory Trait-5 Change Score | Two time point evaluations completed immediately following and 24 hours after biopsy procedure.
  The State Trait Anxiety Inventory Trait-5 (STAIT-5) is a five-item assessment scored on a 4-point Likert scale (1-Not at all, 2-Somewhat, 3-Moderately So, 4-Very Much So) that captures the participants' current state of anxiety with higher scores indicating more anxiety. The five items are as follows: I feel upset, I feel frightened, I feel nervous, I am jittery, I feel confused. The total scores can range from 5 to 20 and the reduction and impact on participants' anxiety while using the Virtual Reality Headset will be based on the change from pre and post biopsy assessments.
Likelihood to Repeat | Single time point evaluation completed 24 hours after biopsy procedure.
  The likelihood of the participant being willing to complete a repeat bone marrow biopsy if deemed medically beneficial will be captured on a 5-point Likert scale immediately following the procedure. Participants will be asked to provide their response to: Please rate your agreement with having the bone marrow biopsy/ bone marrow aspirate procedure done again if deemed medically beneficial. Potential responses can be reported as 1-strongly Disagree, 2-Disagree, 3-Neutral/unsure, 4-Agree and 5-Strongly Agree.

OTHER OUTCOMES:
Number of participants who discontinued study treatment due to adverse events | Evaluation of discontinued study treatment is a periprocedural time point. Estimated time frame is less than 1 hour.
  Specific to the treatment arm only, a binary variable will be determined for each participant indicating whether or not the subject discontinued use of the virtual reality headset due to adverse events (i.e., headache, neck pain, dizziness, seizures, eye strain or muscle twitching, or syncope).

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Varga, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Insitute, Charlotte, North Carolina, United States